CLINICAL TRIAL: NCT07096284
Title: Prognostic Value and Kinetics of the PvCO2-PaCO2/CaO2-CvO2 Ratio Compared to Arterial Lactate in the Initial Phase of Septic Shock
Brief Title: The PvCO2-PaCO2/CaO2-CvO2 Ratio in Septic Shock
Acronym: SepsisO2CO2R
Status: Recruiting | Type: Observational
Sponsor: Avicenna Military Hospital (Other)
Responsible Party: Principal Investigator, Younes Aissaoui, MD, Professor, Avicenna Military Hospital
Other Study IDs: SEPSIS_CO2/O2_vs_lactate
Record Dates: First submitted 2024-12-26; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Septic Shock
Keywords: sepsis; anaerobic metabolism
MeSH Terms: conditions — Shock, Septic; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients with septic shock.: Patients aged over 18 years presenting with septic shock. defined as sepsis with persistent hypotension requiring vasopressors to maintain a mean arterial pressure (MAP) ≥ 65 mmHg and lactatemia > 2 mmol/L despite adequate fluid resuscitation.
  Interventions: Diagnostic Test: PvCO2-PaCO2/CaO2-CvO2 ratio

INTERVENTIONS:
Diagnostic Test: PvCO2-PaCO2/CaO2-CvO2 ratio — Patients diagnosed with septic shock will undergo serial measurements of arterial and venous blood gas analyses, arterial lactate levels, and calculation of the Pv-aCO₂/Ca-vO₂ ratio at predefined time points: H0 (baseline), H2, H6, H12, and H24.
  Calculation Formulas:
  1. Arterial Oxygen Content (CaO₂):CaO2 = SaO2 × Hb × 1,34 + PaO2 × 0,0031
  2. Venous Oxygen Content (CvO₂):CvO2 = SvO2 × Hb × 1,34 + PvO2 × 0,0031
  3. Pv-aCO₂/Ca-vO₂ Ratio: P(v-a) CO2/C(a-v)O2=(PcvCO2-PaCO2)/(CaO2 -CcvO2).

SUMMARY:
The ratio of the venous-arterial carbon dioxide partial pressure difference to the arteriovenous oxygen content difference (Pv-aCO₂/Ca-vO₂) may be a marker of anaerobic metabolism in patients with acute circulatory failure. This study aims to assess the prognostic value of the PvCO2-PaCO2/CaO2-CvO2 in the early phase of septic shock.

DETAILED DESCRIPTION:
The ratio of the venous-arterial carbon dioxide partial pressure difference to the arteriovenous oxygen content difference (Pv-aCO₂/Ca-vO₂) may be a marker of anaerobic metabolism in patients with acute circulatory failure. This study aims to compare the kinetics of the PvCO2-PaCO2/CaO2-CvO2 ratio with a classic marker of anaerobic metabolism (arterial lactate) in the early phase of septic shock.

ELIGIBILITY:
Inclusion Criteria:

Patients aged over 18 years presenting with septic shock, defined as sepsis with persistent hypotension requiring vasopressors to maintain a mean arterial pressure (MAP) ≥ 65 mmHg and lactatemia > 2 mmol/L despite adequate fluid resuscitation. Sepsis is defined by the presence of a suspected or confirmed infectious source associated with organ dysfunction (neurological, respiratory, renal, hepatic, or hematological). [Sepsis 3 criteria]

Exclusion Criteria:

* Absence of central venous access.
* Central venous access not positioned in the superior vena cava (e.g., femoral access).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged over 18 years presenting with septic shock, defined as sepsis with persistent hypotension requiring vasopressors to maintain a mean arterial pressure (MAP) ≥ 65 mmHg and lactatemia > 2 mmol/L despite adequate fluid resuscitation. Sepsis is defined by the presence of a suspected or confirmed infectious source associated with organ dysfunction (neurological, respiratory, renal, hepatic, or hematological). [Sepsis 3 criteria]
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-01-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Prognostic value of PvCO2-PaCO2/Ca O2-CvO2 in patients with septic shock | From patient inclusion (baseilie = H0) then at H2, H6, H 12 and H24 (H = hours)
  The ability of PvCO2-PaCO2/Ca O2-CvO2 to predict mortality in patients with septic shock. These biological values will be measure using arterial and central venous blood gaz.

CONTACTS AND LOCATIONS:
Overall Officials: Younes Aissaoui Pr, Principal Investigator — Cadi Ayyad University. Faculty of Medicine and Pharmacy. Avicenna Military Hospital.
Locations (3):
- Morocco (3):
  - Avicenna Military Hospital, Marrakesh, Marrakesh
  - Avicenna Military Hospital, Marrakesh
  - Department of critical care Medicine. Avicenna Military Hospital, Marrakesh

IPD SHARING:
Plan to Share IPD: Yes
Biological, hemodynamic and outcome data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For 2 years after study completion.

REFERENCES:
- [Result] Ospina-Tascon GA, Madrinan HJ. Combination of O2 and CO2-derived variables to detect tissue hypoxia in the critically ill patient. J Thorac Dis. 2019 Jul;11(Suppl 11):S1544-S1550. doi: 10.21037/jtd.2019.03.52. PMID 31388459